CLINICAL TRIAL: NCT04615221
Title: Immunological Mechanisms of Rejection in Uterine Transplantation
Acronym: MARNI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019_0059
Record Dates: First submitted 2020-10-19; First posted 2020-11-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Graft recipient (Other): During each of the visits carried out with a cervical biopsy as part of the uterine transplant project, samples will be taken.
  Interventions: Other: Specimens
- Living donor (Other): The donors will benefit from a blood sample and a sample of the vaginal microbiota during the transplant under general anesthesia or after it during a consultation scheduled as part of the uterine transplant protocol.
  Interventions: Other: Specimens
- Witness (Other): 10 non-menopausal control patients will each have a cervical biopsy (at different times of the cycle) and a smear, samples of the vaginal microbiota and a blood sample. Among the 10 controls, 4 patients will have to undergo a hysterectomy for which multiple staged biopsies and samples uterine microbiota will be produced.
  Interventions: Other: Specimens

INTERVENTIONS:
Other: Specimens — Specimens (blood, biopsy, cervical smear, vaginal swab)

SUMMARY:
The objective of this study is to understand the mechanisms of rejection in uterine transplantation and to search for non-invasive markers of rejection. The biological samples necessary for our research have been or will be collected during procedures (biopsies, smears, vaginal swab, blood tests) carried out as part of the scheduled follow-up of patients. These will be samples whose collection is minimally or not invasive

DETAILED DESCRIPTION:
In the context of uterine transplantation, non-invasive rejection markers will be sought by different approaches, including transcriptomics on a prospective cohort of patients with different types of samples: blood, smear and biopsy. A microbiota study will also be carried out. 3 groups will be studied: 1 group of 10 patients benefiting or having benefited from a uterine transplant, 1 second group made up of their 10 donors, 1 group of 10 control women

ELIGIBILITY:
Inclusion Criteria:

* Patient going to or having received a uterine transplant OR Patient going to or having donated a uterus for a recipient included in the study OR Premenopausal woman to undergo gynecological surgery under general anesthesia: for 4 of them it was a hysterectomy and they must be under 45 years old, the other 6 must be under 38 years old.

Exclusion Criteria (For witness):

* Pregnancy in progress
* Current infection
* Cervical dysplasia
* History of transplant or transfusion
* Cancer or history of cancer
* Menopause
* Patient aged 38 or over for the 6 controls without hysterectomy, patient aged 45 or over for the 4 patients with hysterectomy.
* Endometriosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
presence of new markers associated with transplant rejection | 8 years

SECONDARY OUTCOMES:
incidence of pregnancy on transplant immunology | 8 years
microbiota in uterine transplant | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Ayoubi, MD, PhD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France